CLINICAL TRIAL: NCT01649674
Title: PRECOL2011-1: Sodium Picophosphate and Magnesium Citrate Versus Polyethylene Glycol as Evacuating Treatment Prior to Colonoscopy: Phase IV Randomized Trial.
Brief Title: Comparison of Bowel Cleansing Regimens Prior to Colonoscopy
Acronym: PRECOL2011-1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRECOL2011-1; 2011-000587-10 (Registry Identifier: EudraCT)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Patients Undergoing Elective Colonoscopy
MeSH Terms: interventions — Solutions; picosulfate sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG (Active Comparator): polyethylene glycol solution 2 liters
  Interventions: Drug: polyethylene glycole (PEG) solution
- NapP (Active Comparator): Sodium picosulphate and magnesium citrate solution 300 ml
  Interventions: Drug: sodium picosulphate and magnesium citrate solution

INTERVENTIONS:
Drug: polyethylene glycole (PEG) solution
  Arms: PEG
Drug: sodium picosulphate and magnesium citrate solution
  Arms: NapP

SUMMARY:
The purpose of this study is to to compare two bowel preparation regimens of patients who will undergo colonoscopy, in terms of quality of bowel preparation and in terms of patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

• Subjects who are candidate to undergo colonoscopy: Diagnosis Screening Follow-up after previous polypectomy

* Informed consent
* Age > 18 years

Exclusion Criteria:

* Previous colonic resection
* Severe inflammatory bowel disease (IBD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2011-11; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale value | at time of colonscopy
  evaluated by two endoscopists who are blinded to treatment assigned at randomization
patient reported acceptability score | just prior to colonscopy
  using visual analog scale

SECONDARY OUTCOMES:
percent of bowel cleansing regimen dose assumed as reported by patient | just prior to colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Valentina D'Angelo, M.D., Principal Investigator — National Cancer Institute, Naples; Mario de Bellis, M.D., Principal Investigator — National Cancer Institute, Naples
Locations (7):
- Italy (7):
  - Presidio Ospedaliero Villa d'Agri, Marsicovetere
  - AO Fatebenefratelli ed Oftalmico, Milan
  - A.O.U. Seconda Universita di Napoli, Napoli
  - Clinica Mediterranea, Napoli
  - Istituto Nazionale dei Tumori, Napoli
  - Presidio Ospedaliero Ascalesi, Napoli
  - Presidio Ospedaliero Maresca, Torre del Greco

REFERENCES:
- [Derived] D'Angelo V, Piccirillo MC, Di Maio M, Gallo C, Bucci C, Civiletti C, Di Girolamo E, Marone P, Rossi GB, Tempesta AM, Tracey MC, Romano M, Miranda A, Taranto D, Sessa G, Esposito P, Salerno R, Pumpo R, De Filippo FR, Della Valle E, de Bellis M, Perrone F. A multicenter randomized phase 4 trial comparing sodium picosulphate plus magnesium citrate vs. polyethylene glycol plus ascorbic acid for bowel preparation before colonoscopy. The PRECOL trial. Front Med (Lausanne). 2022 Dec 8;9:1013804. doi: 10.3389/fmed.2022.1013804. eCollection 2022. PMID 36569131